CLINICAL TRIAL: NCT00293358
Title: SIOP Intracranial Germ Cell Tumours Protocol
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Germ Cell Tumors in the Brain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000455625; CCLG-GC-1997-01; EU-20579; SIOP-CNS-GCT-96
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2008-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood central nervous system germ cell tumor; adult central nervous system germ cell tumor; childhood central nervous system choriocarcinoma; childhood central nervous system embryonal tumor; childhood central nervous system yolk sac tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Carboplatin; Cisplatin; etoposide phosphate; Ifosfamide; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: etoposide phosphate
Drug: ifosfamide
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, etoposide, ifosfamide, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving more than one drug (combination chemotherapy) with radiation therapy may kill more tumor cells.

PURPOSE: This phase III trial is studying combination chemotherapy followed by radiation therapy to see how well it works compared to radiation therapy alone in treating patients with germ cell tumors in the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate and compare, in a non-randomized protocol, reduced-dose craniospinal radiotherapy alone or combination chemotherapy comprising carboplatin, etoposide phosphate, and ifosfamide and local irradiation in patients with intracranial germinoma.
* Increase survival with combination chemotherapy comprising cisplatin, etoposide phosphate, and ifosfamide followed by focal radiotherapy or craniospinal irradiation in patients with intracranial secreting germ cell tumors.

Secondary

* Use the same diagnostic protocol for imaging and laboratory investigations before, during, and after treatment.
* Establish and use a common documentation system regarding general patient's data, including diagnostic tests, clinical evaluation, surgery, histology, radiotherapy, chemotherapy, and toxicity.
* Collect information about toxicity, prognostic factors, and tumor markers.
* Collect epidemiological data, including documentation of incidence and the site and the histologic pattern of intracranial secreting and nonsecreting germ cell tumors in children and adolescents.
* Register associated malformations in the patients as well as the epidemiology of tumors and malformations in relatives.

OUTLINE: This is a non-randomized, multicenter study. Patients are stratified according to tumor classification (pure CNS germinoma vs secreting germ cell tumor and embryonal carcinoma).

Patients in stratum I undergo biopsy or surgical resection and then begin radiotherapy with or without chemotherapy.

* Stratum I (pure CNS germinoma [without elevated markers]): Patients receive 1 of 2 treatment options based on national/center standard:

  * Option 1: Patients receive reduced-dose craniospinal radiotherapy 5 days a week for 3 weeks followed by a boost to the tumor bed 5 days a week for 2 weeks. Patients with multifocal or metastatic disease receive additional boosts to the tumor sites.
  * Option 2: Patients receive carboplatin IV over 1 hour on day 1, etoposide phosphate IV over 1 hour on days 1-3 and 22-24, and ifosfamide IV over 3 hours on days 22-26. Treatment repeats every 6 weeks for 2 courses. After recovery from chemotherapy, patients undergo radiotherapy 5 days a week for 5 weeks.
* Stratum II (secreting tumors and embryonal carcinoma): Patients receive etoposide phosphate IV over 1 hour on days 1-3, cisplatin IV over 1 hour on days 1-5, and ifosfamide IV over 22 hours on days 1-5. Treatment repeats every 3 weeks for up to 4 courses. Patients whose tumor markers do not return to normal after completion of chemotherapy are off protocol. Patients may undergo surgery after chemotherapy course 2 or 4 if required. After completion of chemotherapy and recovery from surgery, patients with nonmetastatic disease undergo radiotherapy to the tumor bed 5 day a week for 6 weeks, and patients with metastatic disease undergo radiotherapy to the cerebrum, spinal axis, and tumor bed for 7 weeks.

After completion of study treatment, patients are followed for 4 weeks and then periodically.

PROJECTED ACCRUAL: Approximately 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinical and radiological evidence of intracranial germ cell tumor, classified as 1 of the following:

  * Germinoma

    * Pure germinoma
    * Germinoma with mature and/or immature teratoma
  * Secreting germ cell tumor

    * Elevated tumor markers in serum and/or cerebral spinal fluid as evidenced by any of the following:

      * Alpha-fetoprotein > 25 ng/mL
      * β-human choriogonadotropin > 50 IU/L
    * Any tumor containing 1 of these components:

      * Yolk sac tumor
      * Choriocarcinoma
      * Embryonal tumor

        * Normal tumor markers allowed
* Diagnosis confirmed by histology or elevated serum markers
* Metastatic or nonmetastatic disease

  * Two separate tumors in the suprasellar and pineal areas without evidence of metastatic disease elsewhere are considered nonmetastatic multifocal disease
* Study treatment must begin ≤ 4 weeks after diagnosis
* No pure immature or mature teratomas
* The following additional patients are eligible:

  * Patients who are > 18 years of age provided no other appropriate protocol exists
  * Patients who were diagnosed > 4 weeks ago
  * Patients who are in relapse

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior treatment except surgery
* No concurrent amino glycosides or other nephrotoxic drugs during ifosfamide administration
* No concurrent growth factors
* No other concurrent chemotherapy or radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 1997-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Survival
Event-free survival

CONTACTS AND LOCATIONS:
Overall Officials: James Nicholson, DM, MA, MRCPCH, Study Chair — Cambridge University Hospitals NHS Foundation Trust; Marie C. Baranzelli, MD — Centre Oscar Lambret; U. Gobel, MD — Heinrich-Heine University, Duesseldorf
Locations (21):
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Derived] Rajagopal R, Leong SH, Jawin V, Foo JC, Ahmad Bahuri NF, Mun KS, Azman RR, Loh J, Yap TY, Ariffin H, Moreira DC, Gottardo NG, Bouffet E, Ganesan D. Challenges in the Management of Childhood Intracranial Germ Cell Tumors in Middle-Income Countries: A 20-Year Retrospective Review From a Single Tertiary Center in Malaysia. J Pediatr Hematol Oncol. 2021 Oct 1;43(7):e913-e923. doi: 10.1097/MPH.0000000000002116. PMID 33633029